



# BPIT Clinical Study Protocol (Version 3.3): Document1

Date: 2025-12-08

Balanced Progressive Intensity Training (BPIT): Multi-Site Clinical Study on Movement Efficiency, Mobility, and Strength Adaptation

**DOI:** 10.5281/zenodo.17594478

ClinicalTrials.gov ID NCT07256717

IMSO: IMSO-REG-20251125-PM-1458-TA

#### **Institutional Header**

MMSx Authority Institute for Movement Mechanics & Biomechanics Research
In Collaboration with BodyGNTX Institute | GFFI India | IIKBS | Bureau of Fitness Standards
(BFS) | Active India Health & Fitness Trust (AIHFT)

| Field | Detail |
|--------------------------|-------------------------------------------------|
| Study Title | Balanced Progressive Intensity Training (BPIT): |
| | A Five-Week Multi-Site Clinical Evaluation of |
| | Functional Movement, Mobility, and |
| | Neuromuscular Adaptation in Healthy Adults |
| | (18-65 years) |
| Principal Investigator | Dr. Neeraj Mehta, Ph.D. (Biomechanics & |
| | Alternative Medicine), Clinical Biomechanics & |
| | Research Ethics Certified (OHRP-HHS USA |
| | ICMR India) |
| Collaborating Institutes | MMSx Authority Institute BodyGNTX GFFI |
| | India IIKBS BFS AIHFT |
| Study Type | Prospective, observational intervention study |
| Study Duration | 5 Weeks |
| Study Sites | BFS- and AIHFT-approved training & |
| | rehabilitation centers |
| IMSO Accreditation ID | [Insert IMSO Accreditation ID] |





## **Version History Section**

Version History:

- Version 3.0: Original draft, July 2025 (anticipated).
- Version 3.1: Minor updates for multi-site details, November 6, 2025.
- Version 3.2: Reviewed for ClinicalTrials.gov submission on November 25, 2025; no substantive changes to study design or methods.
- Version 3.3: Reviewed for ClinicalTrials.gov submission on 2025-12-08; no substantive changes to study design or methods.

## 2. About the BPIT Method (Revised)

Balanced Progressive Intensity Training (BPIT) is a biomechanical and physiological strength-training framework created by Dr. Neeraj Mehta. Its primary goal is to harmonize intensity progression, internal load distribution, and neuromuscular efficiency, thereby resolving the traditional training-injury paradox.

#### 2.1. The BPIT 5-Line Principle

BPIT organizes all strength and movement exercises into five distinct intensity lines. Each line is defined by specific physical parameters, enabling a safe and structured progression from stability to power without generating overuse stress.

| Line | Movement Base | Target HR (bpm) | Focus & Purpose | Examples |
|---|---|---|---|---|
| 1 – | Floor / Low GRF | 95-110 | Core activation + | Plank, Crunch, |
| <b>Ground-Based</b> | | | breath stability | Dead Bug |
| 2 – Knee-Level | Supported /<br>Moderate GRF | 100-120 | controlled press / | Bench Press,<br>Seated Row |
| 3 – Standing | Full Bodyweight | 120-140 | pull Alignment & Kinetic-integration chain | Squat, Deadlift |
| 4 – Head-Level | Overhead /<br>Elevated | 140-160 | Thoracic mobility & scapular control | Overhead Press,<br>Lunge |
| 5 – Plyometric | Dynamic Impact | 160-180 | Elastic power & | Jump Squat, |





| Line | Movement Base | Target HR (bpm) | Focus & Purpose | Examples |
|---|---|---|---|---|
| | | | injury resilience | Burpee, Box Jump |

#### 2.2. Biomechanical Framework

The BPIT methodology operates by balancing **mechanical stimulus \times biomechanical integrity \approx physiological recovery**, ensuring consistent adaptation. Key biomechanical control mechanisms include:

- Ground Reaction Force (GRF) management
- Joint-Load Distribution analysis
- Heart-Rate (HR) and Heart Rate Variability (HRV) Control

#### 3. Study Objectives

- 1. Evaluate the effect of BPIT on movement efficiency, mobility, and load control.
- 2. Quantify biomechanical and neuromuscular changes across the 5-week period.
- 3. Observe individual variance in adaptation and note any mobility or postural deviations.
- 4. Identify early-stage indicators of overload to refine safety parameters.

### 4. Methodology

#### 4.1. Design and Participants

- **Design:** Multi-site, prospective, real-world clinical observation.
- Participants: \geq 369 healthy adults (18-65 years).
- Inclusion Criteria: No acute injury / medically cleared for exercise.
- Exclusion Criteria: Chronic pathology, cardiac instability, recent surgery.
- **Sample size:** n=100 for 80% power (α=0.05, effect size=0.5 via G\*Power 3.1), detecting moderate changes in MES/ROM with 10% dropout.
- Control group: Standard progressive overload training (no BPIT lines) for comparison.
- Additional exclusions: BMI >35, pregnancy, uncontrolled hypertension, or recent surgery (<6 months).

#### 4.2. Procedure: 5-Week Progression





| Week | Phase | Focus | Assessment Tool | Expected |
|---|---|---|---|---|
| | | | | Outcome |
| 0 | Baseline | Posture & Mobility | MMSx Flaw | Establish |
| | Screening | | Checklist + BPIT | Reference |
| | | | Line Mapping | |
| 1-2 | Correction Phase | Stability & Joint | Controlled | \downarrow |
| | | Centration | Low-Load BPIT | Compensation |
| | | | | Patterns |
| 3-4 | Progressive Phase | Load Adaptation & | Mid-Load BPIT | \uparrow MES & |
| | | Efficiency | | ROM |
| 5 | Evaluation Phase | Power Integration | Final BPIT Test + | \uparrow Strength |
| | | | Clinical ROM | & Control |

#### 5. Data Collection Parameters

All data will be stored in the **BodyGNTX Research Registry** with anonymized codes.

| Variable | Metric/Tool | Evaluator | Frequency |
|-----------------------|----------------------|----------------|------------|
| Movement Efficiency | BPIT Observation | MMSx Expert | Weekly |
| Score (MES) | Scale 0-10 | | |
| Range of Motion | Goniometer / Digital | Assessor | Wk 0, 3, 5 |
| (ROM) | Арр | | |
| Pain Scale (VAS 0-10) | Self-Report | Site Clinician | Weekly |
| Strength Index | Rep x Load Chart | Trainer | Wk 0, 5 |
| Postural Symmetry | Video Analysis | Research Staff | Wk 0, 5 |

## 6. Ethical & Medical Oversight

- Study conducted per Declaration of Helsinki (2013) and WHO GCP guidelines.
- Participants must sign the official MMSx Informed Consent Form before initiation.
- Any participant showing adverse change in mobility, movement, or health status will be referred to a medical specialist.
- Oversight is provided by registered orthopedic and sports-medicine doctors under the MMSx Clinical Board.

## 7. Expected Outcomes (Prognosis)





BPIT is projected to validate the model as a safe and scientifically structured progression.

- Movement Efficiency Score improvement by \geq 25\%.
- ROM in major joints improvement by 15-20\%.
- Strength Index improvement by 20-30\%.
- Injury risk reduction by \geq 35\%.

## 8. Signatures

| Role | Name / Institution | Signature | Date |
|---|---|---|---|
| Principal Investigator | Dr. Neeraj Mehta -<br>MMSx Authority | Shupa | 2025-12-08 |
| Site Expert / Clinician | [Name / Institution] | | |
| Medical Observer /<br>Orthopedist | [Name / Institution] | | |
| IRB / Ethics Approval | [MACREB Chair Name] | | |

©2025 MMSx Authority Institute for Movement Mechanics & Biomechanics Research Mehta, N., March. S, . Smith J., & Malhotra, S. (2025). Balanced Progressive Intensity Training (BPIT): A Multi-Site Clinical Evaluation of Movement Efficiency, Mobility, and Strength Adaptation (v3.3) (v3.3) [Data set]. Zenodo. https://doi.org/10.5281/zenodo.17594478